CLINICAL TRIAL: NCT02018744
Title: Multicenter, Observational, Post-Market, Real World Registry to Assess Outcomes of Patients Treated With the Nellix® System for Endovascular Abdominal Aortic Aneurysm Repair
Brief Title: Nellix® Registry Study: EVAS-Global
Acronym: EVAS-FORWARD 1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0010-Ver. 1
Record Dates: First submitted 2013-11-18; First posted 2013-12-23 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Safety and Performance of the Nellix Endovascular Sealing System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry has been designed as a multicenter, single arm, open label, post-market registry study with consecutive, eligible patient enrollment at each site. All subjects undergoing the Endovascular Aneurysm Sealing System (EVAS) with the Nellix®-System. Subjects will be followed up to discharge discharge, and as per institutional standard of care thereafter through to 5 years (total follow-up commitment). This registry of the Nellix System, which has received the market authorization of the European Union (Conformité Européenne, CE-certification) in a "real world" patient population treated in a multicenter setting will provide an assessment of the generalizability of the approach and System.

Up to 300 patients diagnosed with abdominal aortic aneurysm (AAA) who are considered candidates for Endovascular Repair, in up to 30 international centers will be enrolled in the study.

DETAILED DESCRIPTION:
1. Baseline: medical history, physical exams, CT image, bloodwork,
2. Procedure: implantation information
3. Discharge: Physical exam, bloodwork and adverse events, if any
4. Follow-up according to institutional standard through to 5 years including Physical exam, CT image or standard of care imaging eg Doppler Ultrasound, bloodwork and adverse events, if any

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old
2. Subject has signed informed consent for data release
3. Subjects with AAA and eligible for endovascular repair

Exclusion Criteria:

1. Currently participating in another study where primary endpoint has not been reached yet
2. Known allergy to any of the device components
3. Pregnant (females of childbearing potential only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 300 patients diagnosed with AAA who are considered candidates for Endovascular Repair, who meet the study eligibility criteria and sign the Informed consent may be subsequently enrolled in the study
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Immediate procedural technical success | Procedure
  Number of subjects where immediate procedural technical success during procedure was noted
Peri-operative Safety Parameters | Up to 30 days
  Number of subjects with procedural Blood loss >1000mL, Mortality (all-cause), Bowel Ischemia, Paraplegia, Renal Failure, Myocardial Infarction, Respiratory Failure, Stroke
Clinical outcome | Up to 5 years
  Number of subjects with Aneurysm rupture, Conversion to open surgical repair, Endoleak of any type, Clinically significant migration, Aneurysm enlargement through to five years, Secondary endovascular procedures of any type through to five years, Secondary endovascular procedures for (resolution of Endoleak of any type; Device occlusion (due to thrombus or other causes); Device migration AAA sac expansion (>5mm diameter increase); Device defect)

OTHER OUTCOMES:
Device Patency and Integrity | Up to 5 years
  Number of subjects with device patency and integrity throughout the study.
In-hospital evaluations | Discharge
  Evaluation of total amount of polymer fill, total endovascular time, anaesthesia time, fluoroscopy time, contrast volume used, total procedure time, estimated blood loss, incidence of transfusion, time in ICU, time to hospital discharge
Distal Complications | 5 years
  Incidence of distal thrombosis, embolization and iliac stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Andrew Holden, Principal Investigator — Auckland City Hospital; Dr. Michel Reijnen, MD, Principal Investigator — Rijnstate Hospital, Arnhem NL
Locations (19):
- Germany (6):
  - Klinikum Augsburg Klinik für Gefäßchirurgie, Augsburg
  - Universitätsklinikum Düsseldorf Klinik für Gefäß- und Endovaskularchirurgie, Düsseldorf
  - Alfried Krupp Krankenhaus Ruttenscheid, Vascular Centre, Essen
  - Universitätsklinikum Heidelberg Klinik für Gefäßchirurgie Im Neuenheimer Feld, Heidelberg
  - Klinikum Sud Nuernberg, Dept of Vascular Surgery, Nuremberg
  - Klinikum Stuttgart Katharinenen Hospital, Stuttgart
- Pauls Stadins Clinical University Hospital Riga, Riga, Latvia
- Hopital Kirchberg, Dept of Cardio-Vascular, Luxembourg-Kirchberg, Luxembourg
- Netherlands (5):
  - Academisch Medisch Centrum Amsterdam, Department of Surgery, Amsterdam
  - Rijnstate Ziekenhuis, Vasculaire Centrum, Arnhem
  - St Antonius Ziekenhuis, Dept of Vascular Surgery, Nieuwegein
  - Erasmus Medical Centre, Dept of Vascular Surgery, Rotterdam
  - St Elisabeth Ziekenhuis, Dept of Vascular Surgery, Tilburg
- Auckland City Hospital Interventional Radiology, Auckland, New Zealand
- Hospital Hamar, Hamar, Norway
- Sweden (2):
  - Orebro University Hospital, Department of General Surgery, Örebro
  - Karolinska University Hospital, Stockholm
- United Kingdom (2):
  - Addenbrooke's Hospital, Dept of Vascular Surgery, Cambridge
  - St. George's Vascular Institute, London